CLINICAL TRIAL: NCT02626533
Title: Persistent Postoperative Pain and Joint Stiffness After Total Knee Arthroplasty Performed for Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-361
Record Dates: First submitted 2015-12-08; First posted 2015-12-10 (Estimated); Results first posted 2024-07-19 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-02

CONDITIONS: Pain; Joint Stiffness
Keywords: Cytokines
MeSH Terms: conditions — Pain | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, and joint fluid aspirate samples will be collected and stored for analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Total knee arthroplasty patients: Patients undergoing total knee arthroplasty for osteoarthritis are enrolled in the study.
  Blood and joint fluid samples will be obtained from patients. Pain type and severity will be assessed at baseline (enrollment), 4 weeks, 3 months, and 6 months postoperatively.
  Interventions: Procedure: Total Knee Arthroplasty

INTERVENTIONS:
Procedure: Total Knee Arthroplasty — Patients will undergo total unilateral knee arthroplasty for osteoarthritis.

SUMMARY:
Persistent pain and joint stiffness after surgery may interfere with recovery and adversely affect quality of life in up to 40% of patients who have undergone total knee arthroplasty. There is growing evidence that inflammation as well as other medical and psychological factors may be associated with osteoarthritis severity, progression, and associated pain severity. This study aims to identify clinical, biological, and psychological factors that contribute to and predict the development of these complications. Identification of such factors may allow us to target preventative measures to the patients at highest risk of persistent postoperative pain and joint stiffness.

ELIGIBILITY:
Inclusion Criteria:

* Elective primary unilateral total knee arthroplasty
* Osteoarthritis with radiologic evidence of "severe narrowing" and/or "bone on bone" in the affected joint
* Patients of surgeons who have agreed to participate in the study
* Age > 18 years
* American Society of Anesthesiologists (ASA) Physical Status 1-3
* Regional anesthesia
* Epidural patient-controlled analgesia (PCA) for postoperative pain
* Adductor canal block for postoperative pain

Exclusion Criteria:

* Contraindication to regional anesthesia, NSAIDs, dexamethasone or acetaminophen
* Use of general anesthesia
* History of >6 weeks of daily opioid use and/or any use of non-prescribed opioids
* Preoperative oral steroid use in the past 6 months
* Intra-articular steroid injection within one month of scheduled surgery in affected joint
* Non-English speakers
* Pre-existing diagnosis of rheumatic disease or autoimmune disease (e.g. rheumatoid arthritis, psoriatic arthritis, inflammatory bowel disease, multiple sclerosis, Type I diabetes)
* Peri-articular injections or infusions for postoperative pain
* Diagnosis of crystalline arthropathy
* Diagnosis of osteonecrosis
* Active infection or use of antibiotics
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital for Special Surgery patients scheduled to undergo unilateral total knee arthroplasty under regional anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-08-28 (Actual); Study Completion 2018-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meghan Kirksey, MD, PhD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sideris A, Malahias MA, Birch G, Zhong H, Rotundo V, Like BJ, Otero M, Sculco PK, Kirksey M. Identification of biological risk factors for persistent postoperative pain after total knee arthroplasty. Reg Anesth Pain Med. 2022 Mar;47(3):161-166. doi: 10.1136/rapm-2021-102953. Epub 2021 Dec 17. PMID 34921052

RESULTS

PARTICIPANT FLOW:
Groups:
- Total Knee Arthroplasty Patients: Patients undergoing total knee arthroplasty for osteoarthritis are enrolled in the study. Blood and joint fluid samples will be obtained from patients, and questionnaires will be administered to assess pain and stiffness.
  Total Knee Arthroplasty: Patients will undergo total unilateral knee arthroplasty for osteoarthritis.
Period: Overall Study
Arm/Group | Total Knee Arthroplasty Patients
Started | 179
POD 1 Follow up (Participants who were successfully contacted for Post-operative day 1 follow up.) | 162
POD 2 Follow up (Participants who were successfully contacted for post-operative day 2 follow up.) | 162
4 Weeks Post-op (Participants who were successfully contacted for 4 weeks post-operation follow up.) | 162
6 Weeks Post-op (Participants who were successfully contacted for 6 weeks post-operation follow up.) | 162
3 Month Post-op (Participants who were successfully contacted for 3 months post-operation follow up.) | 162
6 Months Post-op (Participants who were successfully contacted for 6 months post-operation follow up.) | 162
Stratified to "Stiff" Group (After completing all study activities/follow up, patients were stratified to the "Stiff" group if they reported a certain score across all questionnaires.) | 32
Stratified to "Non-stiff" Group (After completing all study activities/follow up, patients were stratified to the "Non-stiff" group if they reported a certain score across all questionnaires.) | 130
Completed | 162
Not Completed | 17
Not completed — Protocol Violation | 14
Not completed — Patients were found have meet criteria under the exclusion criterion | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Total Knee Arthroplasty Patients (Stiff); Total Knee Arthroplasty Patients (Non-Stiff): Patients undergoing total knee arthroplasty for osteoarthritis are enrolled in the study. Blood and joint fluid samples will be obtained from patients, and questionnaires will be administered to assess pain and stiffness.
  Total Knee Arthroplasty: Patients will undergo total unilateral knee arthroplasty for osteoarthritis.
  Stiffness was defined as ≤ 95° ROM measured with a goniometer at 6 weeks (± 2 weeks).
- Total: Total of all reporting groups
Arm/Group | Total Knee Arthroplasty Patients (Stiff) | Total Knee Arthroplasty Patients (Non-Stiff) | Total
Number analyzed (Participants) | 32 | 130 | 162
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (8.9) | 67.3 (7.9) | 66.9 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 75 | 92
  Male | 15 | 55 | 70
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 1 | 2
  Black or African American | 4 | 11 | 15
  White | 26 | 116 | 142
  Declined/Unknown | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Presence of Persistent Postoperative Pain Using the Numeric Rating Scale (NRS)
Description: Defined as numeric rating scale (NRS) pain score ≥4 with activity in the operated joint. A lower score is a better outcome. 0 is no pain, and 10 is worst pain imaginable.
Time Frame: 6 months after date of surgery
Population: Some patients lost to follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Total Knee Arthroplasty Patients
Number analyzed (Participants) | 111
Participants | 10

2. Secondary Outcome: Patients Who Experienced Postoperative Joint Stiffness
Description: The number of patients that experienced postoperative joint stiffness, defined as ≤95 degrees range of motion.
Time Frame: 6 weeks after date of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Total Knee Arthroplasty Patients
Number analyzed (Participants) | 162
Participants | 32

3. Secondary Outcome: Postoperative Knee Range of Motion
Description: Range of motion at 6 weeks postoperative. Measured as flexion minus extension. Measured in degrees.
Time Frame: 6 weeks after date of surgery
Population: some patients did not answer the questionnaire
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Total Knee Arthroplasty Patients (Stiff) | Total Knee Arthroplasty Patients (Non-Stiff)
Number analyzed (Participants) | 32 | 130
degrees | 84 (15.6) | 115.3 (8.5)

4. Secondary Outcome: NRS Pain at Rest on POD1
Description: NRS pain at rest on postoperative day 1, measured from 0-10, with 0 being no pain at all to 10 being the worst pain imaginable.
Time Frame: 1 day after surgery
Population: some lost to follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- NRS Pain is >=4 With Activity 6 Months Post-op: Patients whose pain with activity is greater or equal to 4 on the numerical rating scale 6 months following surgery.
- NRS Pain is NOT >4 With Activity 6 Months Post-op: Patients whose pain with activity is less than to 4 on the numerical rating scale 6 months following surgery.
Arm/Group | NRS Pain is >=4 With Activity 6 Months Post-op | NRS Pain is NOT >4 With Activity 6 Months Post-op
Number analyzed (Participants) | 15 | 145
units on a scale | 4.9 (3.6) | 3.2 (2.5)

5. Secondary Outcome: NRS Pain With Movement on POD1
Description: NRS pain with movement on postoperative day 1, measured from 0-10, with 0 being no pain at all to 10 being the worst pain imaginable.
Time Frame: 1 day after surgery
Population: Some patients lost to follow up or did not answer questionnaire.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NRS Pain is >=4 With Activity 6 Months Post-op | NRS Pain is NOT >4 With Activity 6 Months Post-op
Number analyzed (Participants) | 13 | 139
units on a scale | 7.6 (2.8) | 4.9 (2.7)

6. Secondary Outcome: Worst NRS Pain on POD1
Description: Worst NRS pain on postoperative day 1, measured from 0-10, with 0 being no pain at all to 10 being the worst pain imaginable.
Time Frame: 1 day after surgery
Population: Some patients lost to follow up or did not answer questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NRS Pain is >=4 With Activity 6 Months Post-op | NRS Pain is NOT >4 With Activity 6 Months Post-op
Number analyzed (Participants) | 15 | 145
score on a scale | 7.7 (2.6) | 6 (2.7)

7. Secondary Outcome: Least NRS Pain on POD1
Description: Least numerical rating scale (NRS) pain on postoperative day 1, measured from 0-10, with 0 being no pain at all to 10 being the worst pain imaginable.
Time Frame: 1 day after surgery
Population: Some patients lost to follow up or did not answer questionnaire.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NRS Pain is >=4 With Activity 6 Months Post-op | NRS Pain is NOT >4 With Activity 6 Months Post-op
Number analyzed (Participants) | 15 | 145
units on a scale | 1.5 (2.3) | 1.2 (1.7)

8. Secondary Outcome: NRS Pain at Rest on POD2
Description: Numerical rating scale (NRS) pain at rest on postoperative day 2, measured from 0-10, with 0 being no pain at all to 10 being the worst pain imaginable.
Time Frame: 2 days after surgery
Population: Some patients lost to follow up or did not answer questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NRS Pain is >=4 With Activity 6 Months Post-op | NRS Pain is NOT >4 With Activity 6 Months Post-op
Number analyzed (Participants) | 14 | 137
score on a scale | 5.3 (3) | 3.2 (2.2)

9. Secondary Outcome: NRS Pain With Movement on POD2
Description: Numerical rating scale (NRS) pain with movement on postoperative day 2, measured from 0-10, with 0 being no pain at all to 10 being the worst pain imaginable.
Time Frame: 2 days after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NRS Pain is >=4 With Activity 6 Months Post-op | NRS Pain is NOT >4 With Activity 6 Months Post-op
Number analyzed (Participants) | 14 | 137
score on a scale | 7.4 (2.1) | 6.2 (2.2)

10. Secondary Outcome: Worst NRS Pain on POD2
Description: Worst numerical rating scale (NRS) pain on postoperative day 2, measured from 0-10, with 0 being no pain at all to 10 being the worst pain imaginable.
Time Frame: 2 days after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NRS Pain is >=4 With Activity 6 Months Post-op | NRS Pain is NOT >4 With Activity 6 Months Post-op
Number analyzed (Participants) | 14 | 137
score on a scale | 9.1 (1.4) | 7.7 (2)

11. Secondary Outcome: Least NRS Pain on POD2
Description: Least numerical rating scale (NRS) pain on postoperative day 2, measured from 0-10, with 0 being no pain at all to 10 being the worst pain imaginable.
Time Frame: 2 days after surgery
Population: Some patients lost to follow up or did not answer questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NRS Pain is >=4 With Activity 6 Months Post-op | NRS Pain is NOT >4 With Activity 6 Months Post-op
Number analyzed (Participants) | 14 | 137
score on a scale | 3.1 (2.4) | 1.8 (2)

12. Secondary Outcome: NRS Pain at Rest 4 Weeks After Surgery
Description: Numerical rating scale (NRS) pain at rest on 4 weeks postoperative, measured from 0-10, with 0 being no pain at all to 10 being the worst pain imaginable.
Time Frame: 4 weeks after surgery
Population: Some patients lost to follow up or did not answer questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NRS Pain is >=4 With Activity 6 Months Post-op | NRS Pain is NOT >4 With Activity 6 Months Post-op
Number analyzed (Participants) | 14 | 126
score on a scale | 2.9 (2.3) | 2 (1.7)

13. Secondary Outcome: NRS Pain With Movement 4 Weeks After Surgery
Description: Numerical rating scale (NRS) pain with movement on 4 weeks postoperative, measured from 0-10, with 0 being no pain at all to 10 being the worst pain imaginable.
Time Frame: 4 weeks after surgery
Population: Some patients lost to follow up or did not answer questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NRS Pain is >=4 With Activity 6 Months Post-op | NRS Pain is NOT >4 With Activity 6 Months Post-op
Number analyzed (Participants) | 14 | 126
score on a scale | 4.3 (2.9) | 3.3 (2.2)

14. Secondary Outcome: Worst NRS Pain 4 Weeks After Surgery
Description: Worst numerical rating scale (NRS) pain 4 weeks postoperative, measured from 0-10, with 0 being no pain at all to 10 being the worst pain imaginable.
Time Frame: 4 weeks after surgery
Population: Some patients lost to follow up or did not answer questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NRS Pain is >=4 With Activity 6 Months Post-op | NRS Pain is NOT >4 With Activity 6 Months Post-op
Number analyzed (Participants) | 14 | 126
score on a scale | 5.9 (2.2) | 5.4 (2.3)

15. Secondary Outcome: Least NRS Pain 4 Weeks After Surgery
Description: Least numerical rating scale (NRS) pain 4 weeks postoperative, measured from 0-10, with 0 being no pain at all to 10 being the worst pain imaginable.
Time Frame: 4 weeks after surgery
Population: Some patients lost to follow up or did not answer questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NRS Pain is >=4 With Activity 6 Months Post-op | NRS Pain is NOT >4 With Activity 6 Months Post-op
Number analyzed (Participants) | 14 | 126
score on a scale | 1.5 (1.6) | 0.8 (1.3)

16. Secondary Outcome: NRS Pain at Rest 3 Months After Surgery
Description: Numerical rating scale (NRS) pain at rest 3 months postoperative, measured from 0-10, with 0 being no pain at all to 10 being the worst pain imaginable.
Time Frame: 3 months after surgery
Population: Some patients lost to follow up or did not answer questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NRS Pain is >=4 With Activity 6 Months Post-op | NRS Pain is NOT >4 With Activity 6 Months Post-op
Number analyzed (Participants) | 11 | 109
score on a scale | 2.4 (2.8) | 0.8 (1.5)

17. Secondary Outcome: NRS Pain With Movement 3 Months After Surgery
Description: Numerical rating scale (NRS) pain with movement 3 months postoperative, measured from 0-10, with 0 being no pain at all to 10 being the worst pain imaginable.
  The average NRS pain for all participants who completed the survey at 3 months is reported.
Time Frame: 3 months after surgery
Population: Some patients lost to follow up or did not answer questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- NRS Pain is >=4 With Activity 6 Months Post-op: Patients whose pain with activity is greater or equal to 4 on the numerical rating scale 3 months following surgery.
- NRS Pain is NOT >4 With Activity 3 Months Post-op: Patients whose pain with activity is less than to 4 on the numerical rating scale 3 months following surgery.
Arm/Group | NRS Pain is >=4 With Activity 6 Months Post-op | NRS Pain is NOT >4 With Activity 3 Months Post-op
Number analyzed (Participants) | 11 | 109
score on a scale | 3.4 (2.7) | 1.5 (1.9)

18. Secondary Outcome: Worst NRS Pain 3 Months After Surgery
Description: Worst numerical rating scale (NRS) pain 3 months postoperative, measured from 0-10, with 0 being no pain at all to 10 being the worst pain imaginable.
  The average worst NRS pain for all participants who completed the survey at 3 months is reported.
Time Frame: 3 months after date of surgery
Population: Some patients lost to follow up or did not answer questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- NRS Pain is >=4 With Activity 3 Months Post-op: Patients whose pain with activity is greater or equal to 4 on the numerical rating scale 3 months following surgery.
Arm/Group | NRS Pain is >=4 With Activity 3 Months Post-op | NRS Pain is NOT >4 With Activity 3 Months Post-op
Number analyzed (Participants) | 11 | 109
score on a scale | 4.1 (2.5) | 2.3 (2.2)

19. Secondary Outcome: Least NRS Pain 3 Months After Surgery
Description: Least numerical pain rating (NRS) pain 3 months postoperative, measured from 0-10, with 0 being no pain at all to 10 being the worst pain imaginable.
  The average least NRS pain for all participants who completed the survey at 3 months is reported.
Time Frame: 3 months after date of surgery
Population: Some patients lost to follow up or did not answer questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NRS Pain is >=4 With Activity 3 Months Post-op | NRS Pain is NOT >4 With Activity 3 Months Post-op
Number analyzed (Participants) | 11 | 109
score on a scale | 0.8 (1.3) | 0.3 (0.9)

20. Secondary Outcome: NRS Pain at Rest 6 Months After Surgery
Description: NRS pain at rest 6 months postoperative, measured from 0-10, with 0 being no pain at all to 10 being the worst pain imaginable.
  The average NRS pain at rest for all participants who completed the survey at 6 months is reported.
Time Frame: 6 months after date of surgery
Population: Some patients lost to follow up or did not answer questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NRS Pain is >=4 With Activity 6 Months Post-op | NRS Pain is NOT >4 With Activity 6 Months Post-op
Number analyzed (Participants) | 14 | 145
score on a scale | 2.4 (2.4) | 0.4 (0.8)

21. Secondary Outcome: Least NRS Pain 6 Months After Surgery
Description: Least NRS pain 6 months postoperative, measured from 0-10, with 0 being no pain at all to 10 being the worst pain imaginable.
  The average least NRS pain for all participants who completed the survey at 6 months is reported.
Time Frame: 6 months after date of surgery
Population: Some patients lost to follow up or did not answer questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NRS Pain is >=4 With Activity 6 Months Post-op | NRS Pain is NOT >4 With Activity 6 Months Post-op
Number analyzed (Participants) | 14 | 145
score on a scale | 0.7 (1.3) | 0.1 (0.4)

22. Secondary Outcome: Worst NRS Pain 6 Months After Surgery
Description: Least NRS pain 6 months postoperative, measured from 0-10, with 0 being no pain at all to 10 being the worst pain imaginable.
  The average worst NRS pain for all participants who completed the survey at 6 months is reported.
Time Frame: 6 months after date of surgery
Population: Some patients lost to follow up or did not answer questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NRS Pain is >=4 With Activity 6 Months Post-op | NRS Pain is NOT >4 With Activity 6 Months Post-op
Number analyzed (Participants) | 14 | 145
score on a scale | 6.5 (2.4) | 1.4 (1.6)

23. Secondary Outcome: Postoperative Knee Injury and Osteoarthritis Outcome (KOOS) Scores
Description: The Knee Injury and Osteoarthritis Outcome Score (KOOS) is a knee-specific instrument, developed to assess the patients' opinion about their knee and associated problems. The KOOS evaluates both short-term and long-term consequences of knee injury. It holds 42 items in 5 separately scored subscales; Pain, other Symptoms, Function in daily living (ADL), Function in Sport and Recreation (Sport/Rec), and knee-related Quality of Life (QOL). A higher score is a better outcome.
  The score is a percentage score from 0 to 100, 0 representing extreme problems and 100 representing no problems.
  Although collected at different timepoints, the average score for each participant is calculated and then the average score for all patients is reported.
Time Frame: 4 weeks, 3 months, and 6 months after date of surgery
Population: This outcome was measured at three different timepoints (4 weeks, 3 months, and 6 months). Some participants could not be reached for follow-up at certain timepoints, therefore the number of patients analyzed for each timepoint differs.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Total Knee Arthroplasty Patients (Stiff) | Total Knee Arthroplasty Patients (Non-Stiff)
Number analyzed (Participants) | 28 | 115
score on a scale
  KOOS Symptoms 4 weeks | 37 (11) | 32 (12)
  KOOS Quality of Life 4 weeks: number analyzed (Participants) | 17 | 61
  KOOS Quality of Life 4 weeks | 18 (15) | 20 (17)
  KOOS Symptoms 3 month: number analyzed (Participants) | 21 | 99
  KOOS Symptoms 3 month | 32 (14) | 33 (13)
  KOOS Quality of Life 3 month: number analyzed (Participants) | 12 | 52
  KOOS Quality of Life 3 month | 19 (26) | 37 (20)
  KOOS Symptoms 6 month: number analyzed (Participants) | 24 | 96
  KOOS Symptoms 6 month | 34 (15) | 34 (13)
  KOOS Quality of Life 6 month: number analyzed (Participants) | 23 | 95
  KOOS Quality of Life 6 month | 41 (21) | 48 (21)

24. Secondary Outcome: Postoperative painDETECT Scores
Description: PainDETECT is a 9-item self-report screening questionnaire developed to detect NeP in conditions like chronic low back pain. PD-Q measures 7 aspects of the quality of the pain experienced, the chronological pattern (time course), and whether or not the pain radiates.
  It is scored from 0 to 38, with total scores of <12 considered = nociceptive pain, 13-18 = possible NeP, and >19 = >90% likelihood of NeP. A lower score is a better outcome.
  Although measured at multiple time points, the average score for each participant is analyzed, and then the average scores for all participants is calculated and reported.
Time Frame: 4 weeks, 3 months, and 6 months after date of surgery
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NRS Pain is >=4 With Activity 6 Months Post-op | NRS Pain is NOT >4 With Activity 6 Months Post-op
Number analyzed (Participants) | 10 | 91
score on a scale
  4 weeks: number analyzed (Participants) | 6 | 51
  4 weeks | 6.7 (4.1) | 7 (4.3)
  3 months: number analyzed (Participants) | 10 | 84
  3 months | 6.2 (4.5) | 3.5 (4)
  6 months | 4.9 (7) | 1.4 (2.4)

25. Secondary Outcome: Types of Preoperative Medications
Description: Statin, gabapentinoid, anticonvulsant, selective serotonin reuptake inhibitor (SSRI), tricyclic antidepressant, serotonin norepinephrine reuptake inhibitor (SNRI), and opioid and non-opioid pain medications.
Time Frame: Before surgery
Population: some patients did not answer the questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Total Knee Arthroplasty Patients
Number analyzed (Participants) | 173
Participants
  used statins | 73
  used gabapentin | 0
  used anticonvulsants: number analyzed (Participants) | 172
  used anticonvulsants | 4
  used selective serotonin reuptake inhibitors | 20
  used tricyclic antidepressants | 1
  used serotonin-norepinephrine reuptake inhibitors: number analyzed (Participants) | 172
  used serotonin-norepinephrine reuptake inhibitors | 4

ADVERSE EVENTS:
Time Frame: up to 6 months
Arm/Group | Total Knee Arthroplasty Patients
All-Cause Mortality (participants affected / at risk) | 0/162
Serious Adverse Events (participants affected / at risk) | 0/162
Other Adverse Events (participants affected / at risk) | 0/162

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-27): https://cdn.clinicaltrials.gov/large-docs/33/NCT02626533/Prot_SAP_000.pdf